CLINICAL TRIAL: NCT07233941
Title: Neuropsychological Profile Characterization in Patients With Migraine: Cognitive Functioning and Psychological Variables
Acronym: CogMIG
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: CogMIG
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Migraine; Migraine Disease
Keywords: migraine; cognition; cognitive impairment
MeSH Terms: conditions — Migraine Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective is to define the neuropsychological profile of patients with migraine and evaluate its association with: psychological outcome measures (anxiety-depressive symptoms, pain catastrophizing, excessive worry, and coping strategies); the clinical profile of migraine; the prodromal, ictal, or interictal phase of the migraine attack; pharmacological therapy; and detoxification treatment in patients with migraine associated with medication overuse headache.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients aged between 18 and 65 years.
* Diagnosis of migraine according to the International Classification of Headache Disorders (ICHD-3) criteria.
* Patients with a history of migraine for at least one year, to ensure the stability of the condition.
* Stability of ongoing treatment for at least 3 months at baseline.
* Understanding of the Italian language.

Exclusion Criteria:

* Severe medical or psychiatric conditions (depression, schizophrenia, psychosis) documented by specific previous diagnoses.
* A history of alcohol or drug abuse.
* Primary sensory deficits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 65 years who suffer from migraines
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Cognitive functioning | 2 years
  Neuropsychological test scores in migraine patients and proportion of participants with cognitive performance significantly different from age- and education-adjusted normative data.

SECONDARY OUTCOMES:
Cognitive functions and psychological, clinical aspects | 2 years
  Correlation between cognitive performance scores and validated measures of anxiety/depression, pain catastrophizing, worry, coping strategies, headache-related impact and disability, and sleep quality in migraine patients.
Cognitive functions and different pharmacological treatments | 2 years
  Differences in cognitive test performance scores among groups of migraine patients receiving different pharmacological treatments
Cognitive functions and medication overuse headache | 2 years
  Change in cognitive test performance scores from pre-detoxification to post-detoxification treatment in patients with migraine and medication overuse headache.
Cognitive functions in the different phases of migraine | 2 years
  Comparison of cognitive test performance scores between ictal and interictal migraine phases and across different durations of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Danilo A Montisano, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kosinski M, Bayliss MS, Bjorner JB, Ware JE Jr, Garber WH, Batenhorst A, Cady R, Dahlof CG, Dowson A, Tepper S. A six-item short-form survey for measuring headache impact: the HIT-6. Qual Life Res. 2003 Dec;12(8):963-74. doi: 10.1023/a:1026119331193. PMID 14651415
- [Background] D'Amico D, Mosconi P, Genco S, Usai S, Prudenzano AM, Grazzi L, Leone M, Puca FM, Bussone G. The Migraine Disability Assessment (MIDAS) questionnaire: translation and reliability of the Italian version. Cephalalgia. 2001 Dec;21(10):947-52. doi: 10.1046/j.0333-1024.2001.00277.x. PMID 11843865
- [Background] Gil-Gouveia R, Martins IP. Clinical description of attack-related cognitive symptoms in migraine: A systematic review. Cephalalgia. 2018 Jun;38(7):1335-1350. doi: 10.1177/0333102417728250. Epub 2017 Aug 28. PMID 28847155
- [Background] Guerra LK, Rehfeldt IR, Lima MT, Petzl-Erler ML, de Messias IJ. BF and C3 genetic polymorphisms in Kaingang Indians from southern Brazil. Hum Hered. 1992;42(3):153-6. doi: 10.1159/000154058. PMID 1511992
- [Background] Gil-Gouveia R, Oliveira AG, Martins IP. The impact of cognitive symptoms on migraine attack-related disability. Cephalalgia. 2016 Apr;36(5):422-30. doi: 10.1177/0333102415604471. Epub 2015 Sep 8. PMID 26350071
- [Background] Vallesi A. On the utility of the trail making test in migraine with and without aura: a meta-analysis. J Headache Pain. 2020 Jun 3;21(1):63. doi: 10.1186/s10194-020-01137-y. PMID 32493204
- [Background] Pizer JH, Aita SL, Myers MA, Hawley NA, Ikonomou VC, Brasil KM, Hernandez KA, Pettway EC, Owen T, Borgogna NC, Smitherman TA, Hill BD. Neuropsychological Function in Migraine Headaches: An Expanded Comprehensive Multidomain Meta-Analysis. Neurology. 2024 Feb 27;102(4):e208109. doi: 10.1212/WNL.0000000000208109. Epub 2024 Jan 22. PMID 38252898
- [Background] Maleki N, Gollub RL. What Have We Learned From Brain Functional Connectivity Studies in Migraine Headache? Headache. 2016 Mar;56(3):453-61. doi: 10.1111/head.12756. Epub 2016 Feb 29. PMID 26924634
- [Background] Mondini S, Montemurro S, Pucci V, Ravelli A, Signorini M, Arcara G. Global Examination of Mental State: An open tool for the brief evaluation of cognition. Brain Behav. 2022 Aug;12(8):e2710. doi: 10.1002/brb3.2710. Epub 2022 Jul 21. PMID 35861637
- [Background] Stern Y. The concept of cognitive reserve: a catalyst for research. J Clin Exp Neuropsychol. 2003 Aug;25(5):589-93. doi: 10.1076/jcen.25.5.589.14571. No abstract available. PMID 12815497
- [Background] Nucci M, Mapelli D, Mondini S. Cognitive Reserve Index questionnaire (CRIq): a new instrument for measuring cognitive reserve. Aging Clin Exp Res. 2012 Jun;24(3):218-26. doi: 10.3275/7800. Epub 2011 Jun 20. PMID 21691143
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771